CLINICAL TRIAL: NCT01660230
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study of the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of 3K3A-APC, a Recombinant Variant of Human Activated Protein C (APC), in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetics of Single and Multiple Ascending Doses of 3K3A-APC in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZZ Biotech, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ZZ-3K3A-001; 2011-000793-60 (EudraCT Number)
Record Dates: First submitted 2012-07-25; First posted 2012-08-08 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: APC, 3K3A, 3K3A-APC, volunteer, healthy
MeSH Terms: interventions — Sodium Chloride; Water

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- 6 µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 1: 6 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 20 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 30 µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 2: 30 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 90 µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 3: 90 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 180 µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 4: 180 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 360 µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 5: 360 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- TBD µg/kg 3K3A-APC, single-dose (Active Comparator): Cohort 6: TBD (not to exceed 720) µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 90 µg/kg 3K3A-APC, q12h for 5 doses (Active Comparator): Cohort 7: 90 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 180 µg/kg 3K3A-APC, q12h for 5 doses (Active Comparator): Cohort 8: 180 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- 360 µg/kg 3K3A-APC, q12h for 5 doses (Active Comparator): Cohort 9: 360 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- TBD µg/kg 3K3A-APC, q12h for 5 doses (Active Comparator): Cohort 10: TBD (not to exceed 720) µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  Interventions: Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
- Matching Placebo, 0.9% NaCl in water (Placebo Comparator): Cohorts 1-10: 0.9% sodium chloride in water and administered as either 20 mL IV infusion over 15 minutes (Cohort 1), or 100 mL IV infusion over 15 minutes (Cohorts 2-10)
  Interventions: Drug: 0.9% NaCl in water

INTERVENTIONS:
Biological: 3K3A-APC, diluted in 0.9% sodium chloride in water
  Arms: 180 µg/kg 3K3A-APC, q12h for 5 doses; 180 µg/kg 3K3A-APC, single-dose; 30 µg/kg 3K3A-APC, single-dose; 360 µg/kg 3K3A-APC, q12h for 5 doses; 360 µg/kg 3K3A-APC, single-dose; 6 µg/kg 3K3A-APC, single-dose; 90 µg/kg 3K3A-APC, q12h for 5 doses; 90 µg/kg 3K3A-APC, single-dose; TBD µg/kg 3K3A-APC, q12h for 5 doses; TBD µg/kg 3K3A-APC, single-dose
Drug: 0.9% NaCl in water
  Arms: Matching Placebo, 0.9% NaCl in water

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetic profile of single and multiple ascending intravenous doses of 3K3A-APC in healthy adult subjects aged 18-55 years.

DETAILED DESCRIPTION:
This is a single-center, sequential-cohort, double-blind, placebo-controlled, single- and multiple-ascending dose study. Eligible adult subjects will be assigned sequentially to 1 of 10 cohorts, at successively higher single doses, followed by successively higher multiple doses.

Single IV Doses: 5 subjects per cohort, aged 18-55, will be randomized in a 4:1 manner to receive active drug (6, 30, 90, 180, 360, and TBD µg/kg) or to receive matching placebo (Cohorts 1-6).

Multiple IV Doses: 8 subjects per cohort, aged 18-55, will be randomized in a 3:1 manner to receive active drug (90, 180, 360, and TBD µg/kg) or to receive matching placebo every 12 hours for 5 doses (Cohorts 7-10).

Single-Dose Cohorts Subjects receiving a single dose will be confined in a Phase 1 unit for 12 hours prior to dosing, during dosing, and for 24 hours after dosing (Study Day 1-2) for observation and PK sampling. Subjects will return on Study Day 4 (~72 hours after infusion) and Study Day 15 for additional safety evaluations. A 28-Day follow-up phone call will be made to subjects to collect AEs that occur within 28-days of the dose.

Multiple-Dose Cohorts Subjects receiving multiple doses will be confined in a Phase 1 unit for 12 hours prior to dosing through 24 hours following the last dose (Study Day 1-4) for observation and PK sampling. Subjects will return on Study Day 6 (~72 hours after last infusion) and Study Day 15 for additional safety evaluations. A 28-Day follow-up phone call will be made to subjects to collect AEs that occur within 28-days of the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating females
2. Both men and women of child-bearing potential (i.e., not surgically sterile or post-menopausal defined as age > 40 years without menses for ≥ 2 years) must agree to use a barrier method of contraception plus a spermicide throughout the study.
3. Age 18 to 55 years, inclusive
4. Body Mass Index (BMI) of 19 to 30 kg/m2, inclusive (see APPENDIX B)
5. Willing and able to complete all study visits
6. Agreement to abstain from smoking and drinking alcoholic beverages from 48 hours prior to randomization through last Study Day (15)
7. Signed informed consent form (ICF)

Exclusion Criteria:

1. Any medical problem for which the subject is being evaluated and/or treated
2. Activated partial thromboplastin time (aPTT) greater than upper limit of normal (ULN)
3. Platelet count < 125,000 cells/mm3
4. International Normalized Ratio (INR) > 1.3
5. Any other clinically significant abnormalities in laboratory values (chemistries, hematology, coagulation studies, and urinalysis - see APPENDIX C)
6. Clinically significant abnormalities on electrocardiogram (ECG)
7. Positive serum βHCG pregnancy test at screening or on Study Day -1 (for all women, regardless of child-bearing potential)
8. Positive urine drug screen at screening or on Study Day -1 (see APPENDIX C)
9. Positive blood test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody
10. Known family history of bleeding or blood clotting disorders
11. History of bleeding diathesis
12. History of liver disease with ongoing coagulopathy
13. Use of any prescription or non-prescription medications or supplements within 7 days prior to Study Day -1, excluding hormonal contraceptives
14. Use of anticoagulant medication within 14 days prior to Study Day -1
15. Major surgery within 60 days prior to Study Day -1
16. Receipt of an investigational drug within 30 days prior to Study Day -1
17. Donation of blood or plasma within 30 days prior to Study Day -1
18. Any other condition, that in the opinion of the Site Investigator, may adversely affect the safety of the subject, the subject's ability to complete the study, or the outcome of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D Lyden, MD, FAAN, Principal Investigator — Cedars-Sinai Medical Center; Howard Levy, MD, PhD, MMM, Study Director — ZZ Biotech, LLC
Locations (1):
- Privatklinik Leech, Graz, Austria

REFERENCES:
- [Derived] Lyden P, Levy H, Weymer S, Pryor K, Kramer W, Griffin JH, Davis TP, Zlokovic B. Phase 1 safety, tolerability and pharmacokinetics of 3K3A-APC in healthy adult volunteers. Curr Pharm Des. 2013;19(42):7479-85. doi: 10.2174/1381612819666131230131454. PMID 24372304

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 µg/kg 3K3A-APC, Single-dose: Cohort 1: 6 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 20 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 30 µg/kg 3K3A-APC, Single-dose: Cohort 2: 30 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 90 µg/kg 3K3A-APC, Single-dose: Cohort 3: 90 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 180 µg/kg 3K3A-APC, Single-dose: Cohort 4: 180 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 360 µg/kg 3K3A-APC, Single-dose: Cohort 5: 360 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 720 µg/kg 3K3A-APC, Single-dose: Cohort 6: TBD (not to exceed 720) 720 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 540 µg/kg 3K3A-APC, Single-dose: Cohort 6: TBD (not to exceed 720) 540 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 90 µg/kg 3K3A-APC, q12h for 5 Doses: Cohort 7: 90 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 180 µg/kg 3K3A-APC, q12h for 5 Doses: Cohort 8: 180 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 360 µg/kg 3K3A-APC, q12h for 5 Doses: Cohort 9: 360 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  3K3A-APC, diluted in 0.9% sodium chloride in water
- 540 µg/kg 3K3A-APC, q12h for 5 Doses: Cohort 10: 540 µg/kg 3K3A-APC, diluted in 0.9% sodium chloride in water and administered as an 100 mL IV infusion over 15 minutes; given every 12 hours for 5 doses
  3K3A-APC, diluted in 0.9% sodium chloride in water
- Matching Placebo, 0.9% NaCl in Water: Cohorts 1-10: 0.9% sodium chloride in water and administered as either 20 mL IV infusion over 15 minutes (Cohort 1), or 100 mL IV infusion over 15 minutes (Cohorts 2-10)
  0.9% NaCl in water
Period: Overall Study
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Started | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 6 | 6 | 6 | 6 | 14
Completed | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 6 | 6 | 6 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 6 | 6 | 6 | 6 | 14 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.25 (10.59) | 28.50 (9.26) | 23.75 (2.36) | 24.00 (2.58) | 28.25 (10.11) | 36.00 (9.90) | 23.75 (2.75) | 27.00 (3.58) | 24.50 (3.78) | 27.50 (13.00) | 25.67 (5.28) | 29.14 (8.08) | 27.03 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 3 | 0 | 2 | 2 | 2 | 1 | 2 | 4 | 8 | 30
  Male | 1 | 2 | 3 | 1 | 4 | 0 | 2 | 4 | 5 | 4 | 2 | 6 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 4 | 4 | 4 | 4 | 1 | 4 | 6 | 6 | 6 | 5 | 13 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 6 | 6 | 6 | 6 | 14 | 64

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events That Meet Dose-limiting Toxicity Criteria Specified in Protocol.
Time Frame: Day 4 for single-dose cohorts
Population: All 'single-dose' subjects who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 2 | 4 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Adverse Events That Meet Dose-limiting Toxicity Criteria Specified in the Protocol.
Time Frame: Day 6 for multiple-dose cohorts
Population: All 'multiple-dose' subjects who received at least one dose of study treatment.
Measure: Number; unit: participants
Groups:
- Matching Placebo, 0.9% NaCl in Water: Cohorts 7-10: 0.9% sodium chloride in water and administered as 100 mL IV infusion over 15 minutes
  0.9% NaCl in water
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: All 'single-dose' subjects who received at least one dose of study treatment and who have sufficient data for PK analysis and who have not been excluded from analysis for protocol deviations or other study-related events that could impact the calculation or interpretation of the pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
ng/mL |  | 248 (64.1) | 745 (33.2) | 1423 (131) | 3562 (512) | 6115 (522) | 4428 (462) |

4. Secondary Outcome: Time at Which Cmax is Observed (Tmax) for 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour (from start of infusion)
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
hour (from start of infusion) |  | 0.250 [0.250 to 0.250] | 0.250 [0.233 to 0.250] | 0.250 [0.250 to 0.333] | 0.333 [0.250 to 0.333] | 0.250 [0.250 to 0.250] | 0.250 [0.250 to 0.250] |

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Final Time With a Concentration ≥ Limit of Quantitation [AUC(0-t)] for 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h * ng/mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
h * ng/mL |  | 85.8 (33.9) | 327 (31.2) | 615 (101) | 1492 (140) | 3025 (174) | 2156 (176) |

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity [AUC(0-inf)] for 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h * ng/mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
h * ng/mL |  | 114 (31.9) | 374 (31.8) | 664 (112) | 1555 (147) | 3087 (178) | 2226 (188) |

7. Secondary Outcome: Elimination Rate Constant (λz) for 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
L/h |  | 3.45 (0.84) | 2.69 (0.50) | 2.73 (0.47) | 2.50 (0.47) | 1.81 (0.32) | 2.03 (0.32) |

8. Secondary Outcome: Half-life (t1/2) of 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
h |  | 0.208 (0.041) | 0.263 (0.043) | 0.259 (0.045) | 0.285 (0.054) | 0.388 (0.069) | 0.347 (0.049) |

9. Secondary Outcome: Total Clearance (CL) of 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
mL/h |  | 18,556 (4,538) | 18,328 (1,686) | 16,883 (573) | 18,036 (1,558) | 12,081 (535) | 17,285 (1,546) |

10. Secondary Outcome: Volume of Distribution (Vz) of 3K3A-APC by Non-compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 4 | 2 | 4 | 0
mL |  | 5,494 (1,501) | 6,934 (1,173) | 6,727 (944) | 7,412 (1,473) | 6,744 (911) | 8,674 (1,655) |

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of 3K3A-APC by Compartmental Analysis
Description: Single-dose cohorts
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
ng/mL |  | 249 (59.2) | 741 (50.2) | 1300 (111) | 3374 (490) | 5715 (306) | 4489 (654) |

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity [AUC(0-inf)] for 3K3A-APC by Compartmental Analysis
Description: Single-dose cohorts; primary parameters (CL, V) were used to fit the model. Secondary parameters (Cmax, AUC(inf), λz, t1/2) were estimated from the primary parameters.
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h * ng/mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
h * ng/mL |  | 123 (32.0) | 381 (29.6) | 623 (131) | 1615 (142) | 3195 (263) | 2309 (191) |

13. Secondary Outcome: Elimination Rate Constant (λz) for 3K3A-APC by Compartmental Analysis
Description: as for outcome 12
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
L/h |  | 2.85 (0.30) | 2.69 (0.49) | 3.08 (0.65) | 2.96 (0.33) | 2.40 (0.44) | 2.68 (0.49) |

14. Secondary Outcome: Half-life (t1/2) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 12
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
h |  | 0.246 (0.027) | 0.263 (0.043) | 0.232 (0.046) | 0.237 (0.029) | 0.294 (0.054) | 0.264 (0.041) |

15. Secondary Outcome: Total Clearance (CL) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 12
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
mL/h |  | 17,017 (4,163) | 18,016 (1,695) | 17,981 (2,321) | 17,372 (1,700) | 11,693 (807) | 16,665 (1,555) |

16. Secondary Outcome: Volume of Distribution (V) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 12
Time Frame: 0, 5, 10, 15, 20, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 6 and 8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 0 | 4 | 4 | 4 | 4 | 2 | 4 | 0
mL |  | 5967 (1236) | 6831 (1231) | 5931 (726) | 5970 (1194) | 4922 (574) | 6359 (1277) |

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of 3K3A-APC by Compartmental Analysis
Description: Multiple-dose cohorts; primary parameters (CL, V) were used to fit the model. Secondary parameters (Cmax, AUC(inf), λz, t1/2) were estimated from the primary parameters.
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: All 'multiple-dose' subjects who received at least one dose of study treatment and who have sufficient data for PK analysis and who have not been excluded from analysis for protocol deviations or other study-related events that could impact the calculation or interpretation of the pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
ng/mL | 810 (118) | 1447 (135) | 2990 (608) | 5577 (1134) |

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity [AUC(0-inf)] for 3K3A-APC by Compartmental Analysis
Description: as for outcome 17
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h * ng/mL
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
h * ng/mL | 370 (145) | 794 (148) | 1634 (365) | 2750 (512) |

19. Secondary Outcome: Elimination Rate Constant (λz) for 3K3A-APC by Compartmental Analysis
Description: as for outcome 17
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
L/h | 3.87 (1.58) | 2.50 (0.46) | 2.47 (0.20) | 2.83 (0.25) |

20. Secondary Outcome: Half-life (t1/2) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 17
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
h | 0.211 (0.097) | 0.284 (0.044) | 0.282 (0.022) | 0.247 (0.022) |

21. Secondary Outcome: Total Clearance (CL) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 17
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
mL/h | 18,701 (4,797) | 17,177 (2,593) | 14,231 (2,536) | 13,647 (1,584) |

22. Secondary Outcome: Volume of Distribution (V) of 3K3A-APC by Compartmental Analysis
Description: as for outcome 17
Time Frame: 0, 20 minutes and 1 hour post for doses 1 and 5
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 0
mL | 5151 (982) | 6971 (1169) | 5732 (645) | 4873 (828) |

ADVERSE EVENTS:
Time Frame: AEs were reported from the first dose of study drug through 28 Days following the last dose (Day 28 Follow-up visit).
Arm/Group | 6 µg/kg 3K3A-APC, Single-dose | 30 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, Single-dose | 180 µg/kg 3K3A-APC, Single-dose | 360 µg/kg 3K3A-APC, Single-dose | 720 µg/kg 3K3A-APC, Single-dose | 540 µg/kg 3K3A-APC, Single-dose | 90 µg/kg 3K3A-APC, q12h for 5 Doses | 180 µg/kg 3K3A-APC, q12h for 5 Doses | 360 µg/kg 3K3A-APC, q12h for 5 Doses | 540 µg/kg 3K3A-APC, q12h for 5 Doses | Matching Placebo, 0.9% NaCl in Water
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/2 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 0/4 | 1/4 | 3/4 | 2/2 | 4/4 | 5/6 | 2/6 | 6/6 | 5/6 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 µg/kg 3K3A-APC, Single-dose (N=4) | 30 µg/kg 3K3A-APC, Single-dose (N=4) | 90 µg/kg 3K3A-APC, Single-dose (N=4) | 180 µg/kg 3K3A-APC, Single-dose (N=4) | 360 µg/kg 3K3A-APC, Single-dose (N=4) | 720 µg/kg 3K3A-APC, Single-dose (N=2) | 540 µg/kg 3K3A-APC, Single-dose (N=4) | 90 µg/kg 3K3A-APC, q12h for 5 Doses (N=6) | 180 µg/kg 3K3A-APC, q12h for 5 Doses (N=6) | 360 µg/kg 3K3A-APC, q12h for 5 Doses (N=6) | 540 µg/kg 3K3A-APC, q12h for 5 Doses (N=6) | Matching Placebo, 0.9% NaCl in Water (N=14)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 4 (4) | 5 (12) | 2 (10) | 6 (27) | 5 (17) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 3 (5)
Migraine (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Samples were analyzed from 4 treated subjects in the 6 μg/kg dose group, but all values were below the lower limit of quantitation for the assay (75 ng/mL) and therefore no PK analysis could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less